CLINICAL TRIAL: NCT00319709
Title: An Eight-Week, Double-Blind Placebo Controlled, Multicenter Study Evaluating the Efficacy, Safety, Tolerability of a Fixed Dose of SR58611A (350 mg q12) in Elderly Patients With Major Depressive Disorder (MDD)
Brief Title: An Eight-Week Study to Evaluate the Efficacy and Safety of SR58611A in Elderly Patients With Depression
Acronym: ZEPHIR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EFC4846; EudraCT 2005-005597-67
Record Dates: First submitted 2006-04-28; First posted 2006-04-27 (Estimated); Last update posted 2009-03-12 (Estimated); Status verified 2009-03

CONDITIONS: Depressive Disorder
Keywords: depression; antidepressive agents; controlled clinical trial
MeSH Terms: conditions — Depressive Disorder; Depression | interventions — Amibegron hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: SR58611A

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of SR58611A in elderly patients with depression.The primary objective is to evaluate the efficacy of a 700 mg dose of SR58611A compared to placebo in elderly patients with depression. The secondary objectives are to evaluate the safety of SR58611A and to evaluate the efficacy of SR58611A on disability and quality of life in elderly patients with depression.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients or inpatients
* Major Depressive Disorder (MDD) with a recurrent Major Depressive Episode (MDE) according to DSM IV-TR criteria.
* MADRS score equal of above 22.

Exclusion Criteria:

* Patients with a current significant risk of suicide in the investigator's clinical judgment.
* The duration of the current depressive episode is greater than 2 years.
* Patients whose current depressive episode is secondary to a general medical condition
* Patients with a lifetime history according to MINI at screening of:bipolar disorder, psychotic disorder, antisocial personality disorder.
* Patients with a current history according to MINI at screening of anxiety disorders, alcohol dependence or abuse or substance dependence or abuse
* Patients with severe or unstable concomitant medical conditions.
* History of seizures other than a single childhood febrile seizure.
* Patients with abnormal thyroid functioning.
* Patients with clinically significant ECG findings at screening.
* Patients who have taken an investigational drug in the last 3 months prior to screening.
* Any subject who has previously participated in a SR58611A protocol.
* Patients with Mini-Mental State Examination (MMSE) score < 25 at screening.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 288 (Actual)
Dates: Start 2006-04; Primary Completion 2007-04 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
The primary outcome of the study is the change from baseline to Day 56 of treatment in the Hamilton Depression Rating Scale (HAM-D) total score.

SECONDARY OUTCOMES:
The main secondary outcomes are the changes from baseline to Day 56 of treatment in the HAM-D depressed mood item, the Montgomery Asberg Depression Rating Scale total, and the Clinical Global Impression Severity of Illness scores.

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (5):
- Sanofi-Aventis Administrative Office, Sofia, Bulgaria
- Sanofi-Aventis Administrative Office, Helsinki, Finland
- Sanofi-Aventis Administrative Office, Bucharest, Romania
- Sanofi-Aventis Administrative Office, Belgrade, Serbia
- Sanofi-Aventis Administrative Office, Bratislava, Slovakia

REFERENCES:
- See also: Related Info — http://www.sanofi-aventis.com